CLINICAL TRIAL: NCT01470222
Title: The Healthy Weight for Life Program
Acronym: HWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susan Roberts, Senior Scientist, Energy Metabolism Laboratory, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9279
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Overweight; Obesity; Compliance Behavior
Keywords: Worksite; group weight loss; behavioral components
MeSH Terms: conditions — Overweight; Obesity; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Monthly, all-worksite activities will be implemented to raise awareness of healthy nutrition for weight control throughout the worksite. The purpose of the all-worksite activities is: a) to create a supportive worksite-wide atmosphere for the individuals enrolling in the weight loss support group, and b) to provide low-level weight loss support for individuals who wish to prevent weight gain.
  Individuals with eligible weight (defined as BMI ≥ 25 kg/m2) without medical contradictions to weight loss, who wish to join a support group to lose weight, may enroll in the worksite weight control support group that will meet weekly for the first 10 weeks and then monthly until the end of the 6-month intervention
  Interventions: Other: Weight loss intervention
- Control Group (delayed intervention) (Experimental): At the end of the study period, subjects will receive a 2-month structured intervention that will provide all of the resources and materials given to the intervention worksite as well as weight control support groups for employees interested in losing weight.
  Interventions: Other: Weight loss intervention

INTERVENTIONS:
Other: Weight loss intervention — Menu-based recommendations to consume a high fiber, low glycemic load diet with education on nutrition and behavior change.

SUMMARY:
This study is a randomized controlled pilot of a work site weight control intervention. The purpose of the pilot is to obtain preliminary data for future NIH submissions. Four work sites were identified through a multistage recruiting process. Work sites were randomized to either the intervention group, which will receive the intervention immediately following randomization or the control group which will receive a shortened intervention over a 1-month period, 6 months after the active intervention sites have completed their program. The intervention will consist of a variety of activities conducted over a 6 month period, that are overseen by a work site-Tufts oversight group, including the following optional elements: For overweight and obese individuals, regular support groups for weight loss and prevention of weight regain. For all work site employees irrespective of weight, handouts and posted informational resources on healthy eating, monthly lunchtime seminars, and food sampling to facilitate healthy eating patterns for prevention of weight gain.

Basic online assessments on health and nutrition will be carried out at baseline (week 0) and 24 weeks in all work site employees willing to provide information. More detailed online and in-person assessments will be performed throughout the 24-week study period in the weight loss support group participants (intervention sites) and individuals intending to enroll in the support group (control sites).

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign a consent form.
* BMI during screening ≥25 kg/m2 (eligibility for weight loss support group)
* Participants must not have had any surgical procedures influencing weight regulation to include, but not limited to, gastric bypass, other bariatric surgeries, resection of small or large intestine leading to malabsorption, gastric resection for ulcers or cancer, and esophageal resection
* Intention to follow recommended program and complete outcome assessments and requested self-monitoring.
* Obtain a physician's clearance form

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Change from baseline weight to weeks 6, 10, 16, 20, 24.
  Fasting Values

SECONDARY OUTCOMES:
*Fasting lipid panel and blood glucose, and blood pressure. Frequency and intensity of use of intervention components by intervention worksite support group employees and their relation to weight change over time. | *Change from baseline to weeks 10 and 24
  questionnaire measures

CONTACTS AND LOCATIONS:
Overall Officials: Sai Krupa Das, Ph.D., Principal Investigator — Tufts University

REFERENCES:
- [Derived] Batra P, Das SK, Salinardi T, Robinson L, Saltzman E, Scott T, Pittas AG, Roberts SB. Eating behaviors as predictors of weight loss in a 6 month weight loss intervention. Obesity (Silver Spring). 2013 Nov;21(11):2256-63. doi: 10.1002/oby.20404. Epub 2013 Jul 2. PMID 23512619
- [Derived] Salinardi TC, Batra P, Roberts SB, Urban LE, Robinson LM, Pittas AG, Lichtenstein AH, Deckersbach T, Saltzman E, Das SK. Lifestyle intervention reduces body weight and improves cardiometabolic risk factors in worksites. Am J Clin Nutr. 2013 Apr;97(4):667-76. doi: 10.3945/ajcn.112.046995. Epub 2013 Feb 20. PMID 23426035